CLINICAL TRIAL: NCT00001711
Title: Volunteer Scanning on MR
Brief Title: Magnetic Resonance Imaging (MRI) Ofl Volunteers
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 980019; 98-CC-0019
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers; Patients
Keywords: Magnetic Resonance Imaging; Gadolinium; MRA; Diagnostic Tool; Contrast; Natural History; Normal Volunteer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers and Patients: Healthy volunteers and patients age 18 and older.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — scan of healthy volunteers.

SUMMARY:
Magnetic resonance is an imaging technique that uses magnetic fields and radio waves to create images of the body. The technology used in magnetic resonance imaging continues to improve. Advancements in magnetic resonance imaging (MRI) requires researchers to study new techniques in normal volunteers in order to understand how to use them in patients with diseases.

In this study researchers plan to do a variety of diagnostic tests including magnetic resonance imaging on normal volunteers. The studies may involve injections of contrast media, substances injected into the blood of participant that improves the image created by the MRI scanner. The study is not expected to benefit the participants. However, information gathered from the study may be used to improve diagnostic techniques and develop new research studies.

DETAILED DESCRIPTION:
Technical evaluation of magnetic resonance imaging and spectroscopy will be performed on subjects who are eligible and willing to volunteer to have a research MRI performed. These studies may involve the administration of commercially available MR contrast media. Some scans may require inhaled carbogen (95% oxygen and 5% carbon dioxide) and hyperoxia (100% oxygen) as a contrast media. The results will be used to evaluate the performance of various pulse sequences, gradient coils, and rf coils on human subjects and will provide essential ground work for specific patient protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any subject above the age of 18 who is capable of giving informed consent. This study allows for the enrollment of healthy volunteers as well as volunteers with disease for the purpose of continued technical development in a wide variety of conditions.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning implanted metal clips or wires of the type which may concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field. Examples include:

1. Aneurysm clip
2. Implanted neural stimulator
3. Implanted cardiac pacemaker or autodefibrillator
4. Cochlear implant
5. Ocular foreign body (e.g., metal shavings)
6. Any implanted device (pumps, infusion devices, etc)
7. Shrapnel injuries
8. All employees/staff supervised by the Principal Investigator or an Associate Investigator are excluded from participation.

To assess whether subjects are normal eligible to participate, they will be asked to fill out a NIH RADIS MRI Safety questionnaire. Subjects will be excluded if it is deemed that they have a condition which would preclude their use for study related MRI (e.g. paralyzed hemidiaphragm, morbid obesity, claustrophobia etc.) or present unnecessary risks (e.g. pregnancy, surgery of uncertain type, symptoms of pheochromocystoma or insulinoma, etc.). Lactating women and subjects with hemoglobinopathies, asthma, or renal or hepatic disease will be excluded from studies involving the administration of contrast agents.

To assess whether subjects are eligible to participate in a GBCA study, before undergoing a GBCA imaging study, volunteers will be asked whether or not they have received a MRI with contrast at an outside institution within the last 6 months and have their Clinical Center medical records reviewed. To track exposures to intravenous GBCAs, for each subject we are administrating GBCA, we will maintain a database recording any reports of GBCA administration at an outside institution and the running total of GCBA administration at the Clinical Center. Volunteers who have had exposure to intravenous GBCAs within the last 6 months at an outside institution or the Clinical Center, or reached their maximum of 4 GBCA research imaging studies during their study participation on this protocol, will be excluded from having a contrast enhanced MRI, but will not be excluded from the protocol for non-contrasted MRI studies.

To ensure volunteers who have renal failure do not undergo a GBCA imaging study, all volunteers who will receive Gadolinium based contrast agents will have a serum Creatinine obtained within one week of the MRI examination. All subjects with a calculated eGFR less than or equal to 60 will be excluded from having a contrast enhanced MRI, but will not be excluded from the protocol for non-contrasted MRI studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any subject above the age of 18 who is capable of giving informed consent. This study allows for the enrollment of healthy volunteers as well as volunteers with disease for the purpose of continued technical development in a wide variety of conditions.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1229 (Actual)
Dates: Start 1998-02-06 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
To develop and optimize new MR techniques for ultimate use in patient protocols | End of study
  develop and optimize new MR techniques for ultimate use in patient protocols.

CONTACTS AND LOCATIONS:
Overall Officials: John A Butman, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.we are working on deciding if we will share IPDs.

REFERENCES:
- [Background] Choyke PL, Walther MM, Wagner JR, Rayford W, Lyne JC, Linehan WM. Renal cancer: preoperative evaluation with dual-phase three-dimensional MR angiography. Radiology. 1997 Dec;205(3):767-71. doi: 10.1148/radiology.205.3.9393533.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Frank JA, Mattay VS, Duyn J, Sobering G, Barrios FA, Zigun J, Sexton R, Kwok P, Woo J, Moonen C, et al. Measurement of relative cerebral blood volume changes with visual stimulation by 'double-dose' gadopentetate-dimeglumine-enhanced dynamic magnetic resonance imaging. Invest Radiol. 1994 Jun;29 Suppl 2:S157-60. doi: 10.1097/00004424-199406001-00052. No abstract available. PMID 7928216
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1998-CC-0019.html